CLINICAL TRIAL: NCT05507229
Title: A Phase III Randomized, Modified Double-blind, Multi-centric, Comparative Study, to Evaluate the Non-inferiority of Immunogenicity and Safety of Single Strain Oral Cholera Vaccine Hillchol® (BBV131)to the Comparator Vaccine Shanchol™ Along With Lot-to-lot Consistency of Hillchol® (BBV131).
Brief Title: A Phase III Randomized, Modified Double-blind, Multi-centric, Comparative Study, to Evaluate the Non-inferiority of Immunogenicity and Safety of Hillchol® (BBV131)to Shanchol™ Along With Lot-to-lot Consistency of Hillchol®(BBV131).
Acronym: Hillchol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hillchol®BBV131/2021
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Hillchol®(BBV131) vaccine - (Lot-I ) administered to 450 subjects on day 0 and 14.
  Interventions: Biological: Hillchol vaccine
- Arm 2 (Experimental): Hillchol®(BBV131) vaccine - (Lot-II) administered to 450 subjects on day 0 and 14.
  Interventions: Biological: Hillchol vaccine
- Arm 3 (Experimental): Hillchol®(BBV131) vaccine - (Lot-III ) administered to 450 subjects on day 0 and 14 .
  Interventions: Biological: Hillchol vaccine
- Arm 4 (Active Comparator): Shanchol Vaccine administered to 450 subjects on day 0 and 14
  Interventions: Biological: Shanchol Vaccine

INTERVENTIONS:
Biological: Hillchol vaccine — HillChol®(BBV131) (Whole cell inactivated Stable Hikojima expressing both Inaba and Ogawa LPS) inactivated bacteria of a stable recombinant Vibrio cholerae O1 El Tor Hikojima serotype strain expressing approximately 50% each of Ogawa and Inaba O1 LPS antigens.
  Arms: Arm 1; Arm 2; Arm 3
Biological: Shanchol Vaccine — Shanchol™ (Killed Bivalent (O1 and O139) Whole Cell Oral Cholera Vaccine)
  Arms: Arm 4

SUMMARY:
A Phase III randomized, modified double-blind, multi-centric, comparative study, to evaluate the noninferiority of immunogenicity and safety of single strain oral cholera vaccine Hillchol® (BBV131) to the comparator vaccine Shanchol™ along with lot-to-lot consistency of Hillchol® (BBV131).

Study Population: A total of 1800 participants will be enrolled in three descending age groups (Group I- >18, Group II: > 5 to <18 and Group-III: >1 to <5) in 3(1350):1(450) ratio. In each group 600 participants will be enrolled and among 600 participants 450 participants will receive any lot of Hillchol® (BBV131) and 150 participants will receive Shanchol™.

DSMB and report:After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I,10-Lot-II,10-Lot-III and 10-shanchol) in the Group I, safety data of these participants will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group I and starting recruitment of participants for group II.

After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I,10-Lot-II,10-Lot-III and 10-shanchol) in the Group II, safety data of these participants will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group II and starting recruitment of participants for group III.

After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131): 10-Lot-I, 10-Lot-II, 10-Lot-III and 10-shanchol) in the Group III, safety data of these subjects will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group III.

A Final report will be generated, based on the safety and immunogenicity of the oral cholera vaccine (Hillchol®) will be notified to the Data safety monitoring board and Central Drugs Standard Control Organization (CDSCO), India.

DETAILED DESCRIPTION:
A Phase III randomized, modified double-blind, multi-centric, comparative study, to evaluate the noninferiority of immunogenicity and safety of single strain oral cholera vaccine Hillchol® (BBV131) to the comparator vaccine Shanchol™ along with lot-to-lot consistency of Hillchol® (BBV131)

Study Population: A total of 1800 participants will be enrolled in three descending age groups (Group I- >18, Group II: > 5 to <18 and Group-III: >1 to <5) in 3(1350):1(450) ratio. In each group 600 participants will be enrolled and among 600 participants 450 participants will receive any lot of Hillchol® (BBV131) and 150 participants will receive Shanchol™.

Study objectives:

Primary Objectives:

1) To demonstrate non-inferiority of immunogenicity Hillchol®(BBV131) to that of Shanchol by comparing the seroconversion rate (defined as '4 fold rise in vibriocidal antibody titer compared to baseline') upon administration of 2 doses of Hillchol®(BBV131) or Shanchol, across all age groups. Secondary

Secondary objectives:

1. To evaluate and compare the immunogenicity of Hillchol®(BBV131) with that of Shanchol across all age groups, by comparing the geometric mean titers (GMT) of vibriocidal antibodies in participants receiving Hillchol®(BBV131) and ShancholTM.
2. To evaluate and compare the frequency and severity of all solicited and unsolicited adverse events upon administration of two doses of Hillchol®(BBV131) or ShancholTM, among all three age groups.

Exploratory Objectives:

1)To demonstrate the consistency of immunogenicity for 3 consecutive lots of Hillchol®(BBV131) (lot-to-lot consistency) across all age groups, by comparing the GMT of vibriocidal antibodies in participants receiving doses from each vaccine lot of Hillchol®(BBV131).

Study Endpoints/Outcome:

1. The proportion of participants achieving seroconversion against Ogawa serotype, 14 days after 2 doses of test or comparator vaccine.
2. The proportion of participants achieving seroconversion against Inaba serotype, 14 days after 2 doses of test or comparator vaccine.
3. Geometric Mean Titers (GMT) of anti-Ogawa antibodies two weeks after 2 doses of Test or comparator vaccine
4. GMT of anti-Inaba antibodies two weeks after 2 doses of Test or comparator vaccine.
5. Immediate reaction: Within 30 mins of administration of each dose.
6. Incidence, intensity, the causality of all solicited adverse events during the 7-day follow-up period after each dose.
7. Incidence, intensity, the causality of unsolicited adverse events during the 14-day follow-up period after each dose.
8. Incidence, intensity, the causality of all adverse events and Serious Adverse Events (SAEs) during the entire study period.
9. The proportion of participants achieving seroconversion against Ogawa and Inaba serotype, 14 days after 2 doses for each consecutive batch of Hillchol®(BBV131).

Sero-conversion is defined as a 4-fold rise above the baseline 14 days post-second dose Geometric mean of vibriocidal antibody titers to be calculated.

Study design:

In this study, a total sample size of 1800 participants will be enrolled in three groups in age descending manner and administered with Hillchol®(BBV131) or Shanchol™.

A) Group-I (Age :> 18): In this group, a total of 600 participants aged >18 will be enrolled and randomly assigned into 1:1:1:1 ratio to receive either any three lots of Hillchol®(BBV131) (150: Lot-I, 150: Lot-II and 150: Lot-III) or Shanchol® (150) on day 0 and 14.

After completion of 7 days post, 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I, 10-Lot-II,10-Lot-III and 10-shanchol) in the Group I, safety data of these participants will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, the study will progress by recruiting remaining 560 participants in the group I and starting recruitment of participants for group II.

B) Group-II (Age: >5 to <18): In this group, a total of 600 participants aged >5 to <18 will be enrolled and randomly assigned into 1:1:1:1 ratio to receive either any three lots of Hillchol® (BBV131)(150: Lot-I, 150: Lot-II and 150: Lot-III) or Shanchol®(150)on day 0 and 14.

After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I,10-Lot-II,10-Lot-III and 10-shanchol) in the Group II, safety data of these participants will be reviewed by the Data Safety Monitoring Board (DSMB) and based on their recommendation, the study will progress by recruiting remaining 560 participants in the group II and starting recruitment of participants for group III.

C) Group-III (Age: >1 to <5): In this group, a total of 600 participants aged >1 to <5 will be enrolled and randomly assigned into 1:1:1:1 ratio to receive either any three lots of Hillchol® (BBV131) (150: Lot-I, 150: Lot-II and 150: Lot-III) or Shanchol® (150) on day 0 and 14.

After completion of 7 days post, 1st dose for 40 participants (Hillchol (BBV131): 10-Lot-I, 10-Lot-II, 10-Lot-III and 10-shanchol) in the Group III, the safety data of these subjects will be reviewed by the Data Safety Monitoring Board (DSMB) and based on their recommendation, the study will progress by recruiting the remaining 560 participants in the group III.

Eligibility Criteria:

Inclusion Criteria

1. Participants /Legally acceptable representatives who have ability to provide written informed consent.
2. Participants of either gender of age > 1 year.
3. Expressed interest and availability to fulfil the study requirements.

   1. Willing to receive two dosesof the vaccine at the specific study site.
   2. Willing to be contacted on the phone to assess adverse events and for study reminders.
4. Agrees not to participate in another clinical study at any time during the study period.

Exclusion

1. Any history of anaphylaxis in relation to vaccination.
2. Participant with Immune function disorders including immunodeficiency diseases, or taking immunosuppressive/cytotoxic agents.
3. An individual thought to have difficulty participating in the study due to severe chronic diseases, based on the judgment of the investigator.
4. Participants with 38℃ or higher body temperature measured within 24 hours or at the time of investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours prior to study initiation
6. Diarrhea or administration of anti-diarrheal drugs or antibiotics to treat diarrhea within 1 week prior to study initiation.
7. Other vaccination within 4week prior to study initiation.
8. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months prior to study initiation.
9. Participation in another clinical trial.
10. History of cholera vaccinations or history of cholera diarrhea.
11. Pregnancy, lactation or willingness/intention to become pregnant during the study.
12. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
13. History of any psychiatric condition likely to affect participation in the study.
14. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
15. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the study or would render the subject unable to comply with the protocol

Study Procedure:

Visit 1: Baseline (Day 0) If eligible, study participants will attend the OPD for physical, general examination. Blood samples will be drawn prior to vaccination. A study vaccine will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes to record any adverse event. Diary cards will be distributed to all the participants to record the adverse events after vaccination.

Day 1-7: The study participants will be telephonically followed up by the site for the first 7 days to know their current health status.

Visit 2: (Day 14+2) Study participants will return to the OPD for physical, general examination. Blood samples will be collected for immunogenicity test. A study vaccine will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes to record any adverse event. Diary cards will be distributed to all the participants to record the adverse events after vaccination. Day 15-21: The study participants will be telephonically followed up by the site for the first 7 days to know their current health status.

Visit 3: (Day 28+2) Study participants will return to the OPD for physical, general examination. Blood samples will be withdrawn to assess immunogenicity.

Visit 4: (Day 56±7) Study participants will return to the OPD for physical, general examination. Blood samples will be withdrawn to assess immunogenicity.

Visit 5: (Day 90±7) Study participants will return to the OPD for physical, general examination. Blood samples will be withdrawn to assess immunogenicity.

Visit 6: (Day 180±7) Study participants will return to the OPD for physical, general examination. Blood samples will be withdrawn to assess immunogenicity. Safety Monitoring: Subjects will be observed for 30 minutes after vaccination for immediate adverse events.

Active surveillance will be conducted for all participants for 7 days and 14 days after each dose of vaccine to ascertain information on solicited adverse events and unsolicited adverse events ("Reactogenicity").

Unscheduled visits:

If any subject develops any adverse or serious adverse event or concerned about his/her health, they will be advised to visit the study site during the study follow-up period. All unscheduled visits and details of adverse events will be documented in the source document. Concomitant medications, if any, will also be recorded.

DSMB & Final report:

DSMB and report:After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I,10-Lot-II,10-Lot-III and 10-shanchol) in the Group I, safety data of these participants will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group I and starting recruitment of participants for group II.

After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131):10-Lot-I,10-Lot-II,10-Lot-III and 10-shanchol) in the Group II, safety data of these participants will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group II and starting recruitment of participants for group III.

After completion of 7 days post 1st dose for 40 participants (Hillchol (BBV131): 10-Lot-I, 10-Lot-II, 10-Lot-III and 10-shanchol) in the Group III, safety data of these subjects will be reviewed by Data Safety Monitoring Board (DSMB) and based on their recommendation, study will progress by recruiting remaining 560 participants in the group III.

A Final report will be generated, based on the safety and immunogenicity of the oral cholera vaccine (Hillchol®) will be notified to the Data safety monitoring board and Central Drugs Standard Control Organization (CDSCO), India.

ELIGIBILITY:
Inclusion Criteria:

1. Participants /Legally acceptable representatives who have ability to provide written informed consent.
2. Participants of either gender of age > 1 year.
3. Expressed interest and availability to fulfil the study requirements.

   1. Willing to receive two dosesof the vaccine at the specific study site.
   2. Willing to be contacted on the phone to assess adverse events and for study reminders.
4. Agrees not to participate in another clinical study at any time during the study period.

Exclusion Criteria:

1. Any history of anaphylaxis in relation to vaccination.
2. Participant with Immune function disorders including immunodeficiency diseases, or taking immunosuppressive/cytotoxic agents.
3. An individual thought to have difficulty participating in the study due to severe chronic diseases, based on the judgment of the investigator
4. Participants with 38℃ or higher body temperature measured within 24 hours or at the time of investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours prior to study initiation
6. Diarrhea or administration of anti-diarrheal drugs or antibiotics to treat diarrhea within 1 week prior to study initiation.
7. Other vaccination within 4week prior to study initiation.
8. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months prior to study initiation.
9. Participation in another clinical trial.
10. History of cholera vaccinations or history of cholera diarrhea.
11. Pregnancy, lactation or willingness/intention to become pregnant during the study.
12. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
13. History of any psychiatric condition likely to affect participation in the study.
14. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
15. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the study or would render the subject unable to comply with the protocol.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 14 days after 2 doses of test or comparator vaccine
  The proportion of participants achieving seroconversion against Ogawa serotype, 14 days after 2 doses of test or comparator vaccine.
  2)The proportion of participants achieving seroconversion against Inaba serotype, 14 days after 2 doses of test or comparator vaccine.

SECONDARY OUTCOMES:
Secondary Outcome | two weeks after 2 doses of Test or comparator vaccine
  Geometric Mean Titers (GMT) of anti-Ogawa antibodies two weeks after 2 doses of Test or comparator vaccine
Secondary Outcome | two weeks after 2 doses of Test or comparator vaccine.
  GMT of anti-Inaba antibodies two weeks after 2 doses of Test or comparator vaccine.
Secondary Outcome | Within 30 mins of administration of each dose.
  Immediate reaction
Secondary outcome | during the 7-day follow-up period after each dose.
  Incidence, intensity, the causality of all solicited adverse events
Secondary Outcome | during the 14-day follow-up period after each dose.
  Incidence, intensity, the causality of unsolicited adverse events during the 14-day follow-up period after each dose.
Secondary outcome | during the entire study period.
  Incidence, intensity, the causality of all adverse events and Serious Adverse Events (SAEs)
  .
Secondary outcome | 14 days after 2 doses for each consecutive batch of Hillchol®(BBV131
  The proportion of participants achieving sero-conversion against Ogawa and Inaba serotype

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - King George Hospital,Visakhapatnam, Visakhapatnam, Andhra Pradesh
  - All India Institute of Medical Sciences,Patna, Patna, Bihar
  - Aatman Hospital, Ahmedabad, Gujarat
  - Pt BD Sharma,PGIMS/UHS. Rohtak, Rohtak, Haryana
  - Jeevan Rekha Hospital ,Belgaum, Belagavi, Karnataka
  - Khalatkar Hospital, Nagpur, Nagpur, Maharashtra
  - Redkar Hospital and Research center,Goa, Goa, South Goa
  - Indus Hospital, Hyderabad, Telangana
  - Rana Hospital Pvt Ltd ,Gorakhpur, Gorakhpur, Uttar Pradesh
  - Prakhar Hopsital Pvt Ltd,Kanpur, Kanpur, Uttar Pradesh
  - National Institute of Cholera and Enteric Diseases,Kolkata, Kolkata, West Bengal